CLINICAL TRIAL: NCT06759350
Title: Soy Isoflavonates Versus Placebo on Quality of Life in Menopausal Women: Randomized Double-blind Clinical Trial: FLAVOCAV TRIAL
Brief Title: Soy Isoflavonates Versus Placebo on Quality of Life in Menopausal Women
Acronym: FLAVOCAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Titular professor, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGO-UNAH-48-3-2025
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Menopausal Women; Soy Isoflavone Effect; Quality of Life
Keywords: menopause; Menopausal Women; Soy isoflavone effect; Quality of life
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: double-blind, efficacy, parallel-group, superiority, randomized clinical trial.
Who Masked: Participant, Investigator
Masking Description: To eliminate researcher bias, a third research participant will place the capsules containing the soy isoflavonate in one bottle and the placebo in another bottle. The bottles will be labeled as group A and group B, but the researchers will not know which is in which group, to ensure that the study intervention and the control/placebo are as indistinguishable as possible to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 2 capsules containing 10 mg natural tocotrienols, 40 mg soy isoflavonoids, 540 mg calcium, vitamin D IU.
  Interventions: Dietary Supplement: Soy isoflavone supplement
- control (Placebo Comparator): 2 placebo capsules containing a multivitamin compound.
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Dietary Supplement: Soy isoflavone supplement — 2 capsules containing 10 mg natural tocotrienols, 40 mg soy isoflavonoids, 540 mg calcium, vitamin D IU.
  Arms: Intervention
Other: Control (placebo) group — 2 placebo capsules containing a multivitamin compound.
  Other Names: Multivitamin compound
  Arms: control

SUMMARY:
Within the context of the proposed research study, the effect of soy isoflavonoid supplements on the quality of life and coagulation of menopausal women. It has been observed that menopause, as a physiological process, is associated with alterations in the physical, mental and sexual quality of life, making the use of hormone replacement therapy necessary; however, hormone therapy is associated with hypercoagulability, since it has been seen that women have higher levels of thrombogenic microvesicles such as: platelets with a greater probability of causing blood clotting were more likely to present a greater amount of white matter hyperintensities, which appear in the MRI scan.

DETAILED DESCRIPTION:
The following study is aimed at clarifying the effects of soy isoflavonate supplements on the quality of life and markers of hypercoagulability in menopausal women. The reasons for conducting this research arise from the concern of minimizing side effects such as hypercoagulation caused by hormone replacement therapy, which is intended to be replaced with soy isoflavonates to evaluate its efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Submission of a signed and dated informed consent form.
* Declared willingness to comply with all study procedures and availability for the duration of the study.
* Can read and write
* Female, age 45 to 65 years
* Female with more than 1 year of amenorrhea.
* No hormone replacement therapy or herbal medications in the 6 months prior to the investigation.
* Ability to take oral medication and willing to comply with the <study intervention regimen.
* Agreement to comply with Lifestyle Considerations for the duration of the study.
* Have a smartphone-type cell phone
* Residence in Francisco Morazán

Exclusion Criteria:

* Patient does not sign informed consent
* Patient does not wish to participate
* History of thrombo embolism
* History of cardiovascular disease
* Presence of estrogen-dependent neoplasm
* Presence of abnormal genital bleeding
* Uncontrolled metabolic diseases
* Smoking and drinking habits
* Use of anticoagulant or acetylsalicylic acid
* Known allergic reactions to soy isoflavonate components
* History of thrombophilias such as: Antithrombin deficiency, Protein C deficiency, Protein S deficiency, Factor V Leiden, Prothrombin G20210A, Hyperhomocysteinemia, Antiphospholipid syndrome, Acquired activated protein C resistance.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
MENCAV | One month from the first intervention until 6 months
  Change in MENCAV questionnaire scores, with 37 items likert type scale, the lowest point is zero and the maximun is 259 points

SECONDARY OUTCOMES:
D-dimer | One month from the first intervention until 6 months
  Changes in D-dimer values
side effects | One month from the first intervention until 6 months
  incidence of side effects of soy isoflavones.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc, Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, FM, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Chen LR, Chen KH. Utilization of Isoflavones in Soybeans for Women with Menopausal Syndrome: An Overview. Int J Mol Sci. 2021 Mar 22;22(6):3212. doi: 10.3390/ijms22063212. PMID 33809928